CLINICAL TRIAL: NCT05082818
Title: Outcome of Treating Urinary Bladder Cancer in Sohag University Hospital Between 2016 to 2020
Brief Title: Outcome of Treating Bladder Cancer in Sohag University Hospital
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Refat Ahmed, resident of clinical oncology faculty of medicine Sohag University, Sohag University
Other Study IDs: Soh-Med-21-10-16
Record Dates: First submitted 2021-10-15; First posted 2021-10-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Drug Therapy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Chemotherapy, Radiotherapy and surgery — Trans urethral resection of the tumour or radical cystectomy

SUMMARY:
Retrospective study of outcome of urinary bladder cancer treated in Sohag University hospital in the past 5 years from 2016 to 2020

DETAILED DESCRIPTION:
This study asses the risk factors, prognosis,disease free survival and overall survive rate of treating urinary badder cancer

ELIGIBILITY:
Inclusion Criteria:

* all stages and grades of urinary bladder cancer Any histological types of urinary bladder cancer

Exclusion Criteria:

* presence of other malignancies

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients of both sex and aged from 18 to 80 years old
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 2 weeks after treatment to the time of relapse
  Time from the end of treatment to the date of first relapse

CONTACTS AND LOCATIONS:
Overall Officials: Samah Refaat, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided